CLINICAL TRIAL: NCT04964648
Title: The Validity of Shear Wave Elastography in Diagnosis of Inflammatory and Malignant Pancreatic Diseases
Brief Title: Shear Wave Elastography in Diagnosis of Inflammatory and Malignant Pancreatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ZRMohamed, assistant lecturer, Assiut University
Other Study IDs: SW-EG in pancreatic diseases
Record Dates: First submitted 2021-07-03; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Shear Wave Elastography; Pancreatic Diseases
Keywords: shear wave elastography; pancreatic diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inflammatory pancreatic lesions: older than 18 years with a diagnosis of acute or chronic pancreatitis
  Interventions: Device: shear wave elastography
- Malignant pancreatic lesions: older than 18 years with a diagnosis of pancreatic neoplasm
  Interventions: Device: shear wave elastography
- Control group: Healthy adult subjects
  Interventions: Device: shear wave elastography

INTERVENTIONS:
Device: shear wave elastography — Shear wave elastography (SW-EG), a form of ultrasound elastography used in transabdominal ultrasonography, can measure tissue elasticity by generating shear waves inside the organ using the acoustic radiation force impulse (ARFI) The ultrasound machine monitors shear wave propagation and measures the velocity. The shear wave velocity, displayed in kilopascals (kPa) or meters per second

SUMMARY:
Only a few studies that have assessed the normal range value for pancreatic stiffness, inflammatory and malignant pancreatic lesions, shear wave velocities of healthy parenchyma, acute and chronic pancreatitis, malignant lesions of the pancreas will be evaluated and compared with other conventional imaging modalities, and evaluate its role in assessment of severity and prediction of clinical course/ outcome in patients with inflammatory pancreatic diseases.

DETAILED DESCRIPTION:
The pancreas is a retroperitoneal organ that has several serious inflammatory and malignant diseases can occur, inflammatory diseases include acute and chronic pancreatitis (Janssen et al., 2007).

Acute pancreatitis (AP) is one of the most frequent gastrointestinal causes for hospital admission in the US.

Chronic pancreatitis, although lower in incidence, significantly reduces patients' quality of life (yadav et al., 2013).

Pancreatic cancer has high mortality and is 1 of the top 5 causes of death from cancer. The burden of pancreatic disorders is expected to increase over time (yadav et al., 2013).

AP is an inflammatory condition of the pancreas presenting as abdominal pain and increased levels of pancreatic enzymes in the blood, most commonly caused by bile stones or excessive use of alcohol (Leppäniemi et al., 2019).

It has been associated with significant morbidity, mortality, and hospitalization costs (Janisch et al., 2016).

AP is a common disorder that leads to large number of admissions in Egypt and elsewhere in the world (Ahmed et al., 2016). The overall prevalence rate is 45.1 per 100,000 population (satoh et al., 2011). The severe form comprising about 20-30% of the patients with hospital mortality rates of about 15% (van santvoort et al., 2011).

Chronic pancreatitis (CP) is an inflammatory pancreatic disease characterized by pancreatic infiltration with inflammatory cells, progressive fibrosis, and loss of pancreatic parenchymal tissue (Ito et al., 2015). The global pooled incidence of CP is 40-50 per 100,000 general population per year (Xiao et al., 2016).

The diagnosis of CP is mainly based on the demonstration of the morphological and/or functional changes that develop during the course of the disease. CP is sometimes diagnosed at the progressed stage because no standard diagnostic criteria or method of diagnosing CP at an early stage has been established (Stevens et al., 2010).

As regard neoplastic lesions of pancreas, the global annual incidence rate for pancreas cancer is about 8/100,000 persons. Adenocarcinoma is the most frequent type of pancreatic cancer (Raimondi et al., 2009).

The overall age-adjusted pancreatic cancer mortality rate in Egypt was 1.47/100,000 population (Soliman et al., 2006).

The diagnosis of pancreatic pathology based on a combination of clinical signs and symptoms, imaging techniques and laboratory investigations (Lippi et al., 2012).

Imaging provides a significant contribution to the diagnosis as well as to the assessment of disease severity in patients with inflammatory pancreatic lesions, also can assess the neoplastic pancreatic lesions with accurate detection of extension and follow up of chemotherapeutic effects and survival prognosis (D'Onofrio et al., 2010; Lippi et al., 2012).

Imaging techniques for pancreatic diseases include ultrasound (US) B-mode, contrast enhanced computed tomography (CECT), magnetic resonance imaging (MRI), secretin-magnetic resonance cholangiopancreatography (S-MRCP), endoscopic ultrasonography (EUS), and endoscopic retrograde cholangiopancreatography (ERCP).

All the techniques have variable sensitivity and specificity, with certain disadvantages (Mateen et al., 2012).

Ultrasound B-mode (US) is effective in detection of etiological causes including presence of gallstones, common bile duct calculi, pseudocysts, pseudoaneurysm, and guiding percutaneous aspiration during the follow-up US also depicts the secondary signs for diagnosis of chronic pancreatitis like calcification and dilatation of pancreatic ducts (Munsell et al., 2010).

CECT is more accurate following the onset of acute pancreatitis in assessment and quantification of necrosis. Although MRI is superior to CECT in this respect, however CECT is less expensive and readily available (Mateen et al., 2012).

Typical CECT findings in acute pancreatitis include focal or diffuse enlargement of the pancreas, heterogeneous enhancement with irregular contour of the margins, increased density of peripancreatic fat planes, as well as the presence of intraperitoneal or retroperitoneal fluid collections (Lippi et al., 2012).

There's increasing use of ultrasound elastography for measuring tissue elasticity (hardness).

Shear wave elastography (SW-EG), a form of ultrasound elastography used in transabdominal ultrasonography, can measure tissue elasticity by generating shear waves inside the organ using the acoustic radiation force impulse (ARFI) (Hirooka et al., 2015; Kuwahara et al., 2016).

The ultrasound machine monitors shear wave propagation and measures the velocity. The shear wave velocity, displayed in kilopascals (kPa) or meters per second (Hirooka et al., 2015; Kuwahara et al., 2016).

Using ARFI, qualitative and quantitative determination of the tissue stiffness can be obtained (Bamber et al., 2013).

Qualitative assessment through generation of elastogram (gray scale or red-green-blue) map in which hard tissue areas are shown in black or dark blue, soft tissue areas in white or red and intermediate stiffness tissues are characterized by a yellow/green color indicator. There is no absolute scale of tissue stiffness (Göya et al., 2014).

Quantitative assessment generates numerical value related to the stiffness of tissue within the region of interest (Rees, 2008).

SW-EG is effective for the non-invasive assessment of liver fibrosis in patients with HCV infection especially in advanced stages (F3 and F4) (Moustafa et al., 2017) However, studies on the role of shear wave in a deep-seated organ like pancreas are limited (Hiroki et al., 2009; D'Onofrio et al., 2009).

Galloti et al. (2010) recorded normal values of shear-wave speed for healthy pancreas to be 1.40 m/s.

Another researcher group compared the diagnostic success of shear wave elastography with B-mode ultrasound and CT scan in patients with AP (Bollen et al., 2012).

They found that when using a cut-off value of 1.63 m/s, the sensitivity and specificity of VTQ for the diagnosis of AP were 100% and 98%, respectively (Bollen et al., 2012).

Also, D'Onofrio et al. (2009) diagnosed pancreatic cystadenoma, which mimicked a solid neoplasm at conventional imaging (US and CT), as cystic at shear wave imaging .

Kuwahara et al. (2018) stated that chronic pancreatitis may be diagnosed noninvasively and objectively using SW-EG without performing EUS.

Only a few studies that have assessed the normal range value for pancreatic stiffness, inflammatory and malignant pancreatic lesions; from this point of view, shear wave velocities of healthy parenchyma, acute and chronic pancreatitis, malignant lesions of the pancreas will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Inflammatory pancreatic lesions (acute or chronic pancreatitis)
2. Malignant pancreatic lesions
3. Healthy adult control

Exclusion Criteria:

1. Patient with difficult visualization of the pancreas on B-mode sonography.
2. Patients with acute liver diseases.
3. Obese patient (body mass index >30 kg/m2).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Inflammatory and Malignant pancreatic lesions who will be admitted in Al-Rajhi University Liver Hospital, Assiut, Egypt.
  * control group: Healthy adult subjects who will be evaluated for annual check-up in Al-Rajhi University Liver Hospital, Assiut, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-10 (Estimated); Primary Completion 2022-07-10 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
shear wave elastography (SWE) in diagnosis of inflammatory and malignant pancreatic diseases | Baseline
  •To measure the shear wave velocity (displayed in kilopascals (kPa) or meters per second) of inflammatory and malignant pancreatic diseases
•To compare the diagnostic success rate of shear wave elastography with other conventional imaging modalities | Baseline
  •To compare the diagnostic success rate of shear wave elastography with those of sonography and computed tomography (CT) for inflammatory and malignant pancreatic diseases.

REFERENCES:
- [Background] Bamber J, Cosgrove D, Dietrich CF, Fromageau J, Bojunga J, Calliada F, Cantisani V, Correas JM, D'Onofrio M, Drakonaki EE, Fink M, Friedrich-Rust M, Gilja OH, Havre RF, Jenssen C, Klauser AS, Ohlinger R, Saftoiu A, Schaefer F, Sporea I, Piscaglia F. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 1: Basic principles and technology. Ultraschall Med. 2013 Apr;34(2):169-84. doi: 10.1055/s-0033-1335205. Epub 2013 Apr 4. PMID 23558397
- [Background] Bollen TL, Singh VK, Maurer R, Repas K, van Es HW, Banks PA, Mortele KJ. A comparative evaluation of radiologic and clinical scoring systems in the early prediction of severity in acute pancreatitis. Am J Gastroenterol. 2012 Apr;107(4):612-9. doi: 10.1038/ajg.2011.438. Epub 2011 Dec 20. PMID 22186977
- [Background] D'Onofrio M, Gallotti A, Martone E, Pozzi Mucelli R. Solid appearance of pancreatic serous cystadenoma diagnosed as cystic at ultrasound acoustic radiation force impulse imaging. JOP. 2009 Sep 4;10(5):543-6. PMID 19734634
- [Background] D'Onofrio M, Gallotti A, Pozzi Mucelli R. Imaging techniques in pancreatic tumors. Expert Rev Med Devices. 2010 Mar;7(2):257-73. doi: 10.1586/erd.09.67. PMID 20214430
- [Background] Moustafa EF, Makhlouf N, Hassany SM, Helmy A, Nasr A, Othman M, Seif H, Darwish M, Hassan H, Hessen M. Non-invasive assessment of liver fibrosis in patients with hepatitis C: Shear wave elastography and colour Doppler velocity profile technique versus liver biopsy. Arab J Gastroenterol. 2017 Mar;18(1):6-12. doi: 10.1016/j.ajg.2017.01.004. Epub 2017 Mar 3. PMID 28262531
- [Background] Friedrich-Rust M, Romen D, Vermehren J, Kriener S, Sadet D, Herrmann E, Zeuzem S, Bojunga J. Acoustic radiation force impulse-imaging and transient elastography for non-invasive assessment of liver fibrosis and steatosis in NAFLD. Eur J Radiol. 2012 Mar;81(3):e325-31. doi: 10.1016/j.ejrad.2011.10.029. Epub 2011 Nov 26. PMID 22119555
- [Background] Friedrich-Rust M, Wunder K, Kriener S, Sotoudeh F, Richter S, Bojunga J, Herrmann E, Poynard T, Dietrich CF, Vermehren J, Zeuzem S, Sarrazin C. Liver fibrosis in viral hepatitis: noninvasive assessment with acoustic radiation force impulse imaging versus transient elastography. Radiology. 2009 Aug;252(2):595-604. doi: 10.1148/radiol.2523081928. PMID 19703889
- [Background] Gallotti A, D'Onofrio M, Pozzi Mucelli R. Acoustic Radiation Force Impulse (ARFI) technique in ultrasound with Virtual Touch tissue quantification of the upper abdomen. Radiol Med. 2010 Sep;115(6):889-97. doi: 10.1007/s11547-010-0504-5. Epub 2010 Jan 15. English, Italian. PMID 20082227
- [Background] Goertz RS, Schuderer J, Strobel D, Pfeifer L, Neurath MF, Wildner D. Acoustic radiation force impulse shear wave elastography (ARFI) of acute and chronic pancreatitis and pancreatic tumor. Eur J Radiol. 2016 Dec;85(12):2211-2216. doi: 10.1016/j.ejrad.2016.10.019. Epub 2016 Oct 18. PMID 27842669
- [Background] Goya C, Hamidi C, Hattapoglu S, Cetincakmak MG, Teke M, Degirmenci MS, Kaya M, Bilici A. Use of acoustic radiation force impulse elastography to diagnose acute pancreatitis at hospital admission: comparison with sonography and computed tomography. J Ultrasound Med. 2014 Aug;33(8):1453-60. doi: 10.7863/ultra.33.8.1453. PMID 25063411
- [Background] Uchida H, Hirooka Y, Itoh A, Kawashima H, Hara K, Nonogaki K, Kasugai T, Ohno E, Ohmiya N, Niwa Y, Katano Y, Ishigami M, Goto H. Feasibility of tissue elastography using transcutaneous ultrasonography for the diagnosis of pancreatic diseases. Pancreas. 2009 Jan;38(1):17-22. doi: 10.1097/MPA.0b013e318184db78. PMID 18695627
- [Background] Hirooka Y, Kuwahara T, Irisawa A, Itokawa F, Uchida H, Sasahira N, Kawada N, Itoh Y, Shiina T. JSUM ultrasound elastography practice guidelines: pancreas. J Med Ultrason (2001). 2015 Apr;42(2):151-74. doi: 10.1007/s10396-014-0571-7. Epub 2014 Oct 8. PMID 26576568
- [Background] Ito T, Ishiguro H, Ohara H, Kamisawa T, Sakagami J, Sata N, Takeyama Y, Hirota M, Miyakawa H, Igarashi H, Lee L, Fujiyama T, Hijioka M, Ueda K, Tachibana Y, Sogame Y, Yasuda H, Kato R, Kataoka K, Shiratori K, Sugiyama M, Okazaki K, Kawa S, Tando Y, Kinoshita Y, Watanabe M, Shimosegawa T. Evidence-based clinical practice guidelines for chronic pancreatitis 2015. J Gastroenterol. 2016 Feb;51(2):85-92. doi: 10.1007/s00535-015-1149-x. Epub 2016 Jan 4. PMID 26725837
- [Background] Janisch NH, Gardner TB. Advances in Management of Acute Pancreatitis. Gastroenterol Clin North Am. 2016 Mar;45(1):1-8. doi: 10.1016/j.gtc.2015.10.004. Epub 2015 Dec 19. PMID 26895677
- [Background] Janssen J, Schlorer E, Greiner L. EUS elastography of the pancreas: feasibility and pattern description of the normal pancreas, chronic pancreatitis, and focal pancreatic lesions. Gastrointest Endosc. 2007 Jun;65(7):971-8. doi: 10.1016/j.gie.2006.12.057. PMID 17531630
- [Background] Kaya M, Degirmenci S, Goya C, Tuncel ET, Ucmak F, Kaplan MA. The importance of acoustic radiation force impulse (ARFI) elastography in the diagnosis and clinical course of acute pancreatitis. Turk J Gastroenterol. 2018 May;29(3):342-347. doi: 10.5152/tjg.2018.17338. PMID 29755019
- [Background] Kuwahara T, Hirooka Y, Kawashima H, Ohno E, Sugimoto H, Hayashi D, Morishima T, Kawai M, Suhara H, Takeyama T, Yamamura T, Funasaka K, Nakamura M, Miyahara R, Watanabe O, Ishigami M, Shimoyama Y, Nakamura S, Hashimoto S, Goto H. Quantitative evaluation of pancreatic tumor fibrosis using shear wave elastography. Pancreatology. 2016 Nov-Dec;16(6):1063-1068. doi: 10.1016/j.pan.2016.09.012. Epub 2016 Sep 23. PMID 27692969
- [Background] Kuwahara T, Hirooka Y, Kawashima H, Ohno E, Ishikawa T, Yamamura T, Furukawa K, Funasaka K, Nakamura M, Miyahara R, Watanabe O, Ishigami M, Hashimoto S, Goto H. Usefulness of shear wave elastography as a quantitative diagnosis of chronic pancreatitis. J Gastroenterol Hepatol. 2018 Mar;33(3):756-761. doi: 10.1111/jgh.13926. PMID 28833507
- [Background] Leppaniemi A, Tolonen M, Tarasconi A, Segovia-Lohse H, Gamberini E, Kirkpatrick AW, Ball CG, Parry N, Sartelli M, Wolbrink D, van Goor H, Baiocchi G, Ansaloni L, Biffl W, Coccolini F, Di Saverio S, Kluger Y, Moore E, Catena F. 2019 WSES guidelines for the management of severe acute pancreatitis. World J Emerg Surg. 2019 Jun 13;14:27. doi: 10.1186/s13017-019-0247-0. eCollection 2019. PMID 31210778
- [Background] Lippi G, Valentino M, Cervellin G. Laboratory diagnosis of acute pancreatitis: in search of the Holy Grail. Crit Rev Clin Lab Sci. 2012 Jan-Feb;49(1):18-31. doi: 10.3109/10408363.2012.658354. PMID 22339380
- [Background] Mateen MA, Muheet KA, Mohan RJ, Rao PN, Majaz HM, Rao GV, Reddy DN. Evaluation of ultrasound based acoustic radiation force impulse (ARFI) and eSie touch sonoelastography for diagnosis of inflammatory pancreatic diseases. JOP. 2012 Jan 10;13(1):36-44. PMID 22233945
- [Background] Munsell MA, Buscaglia JM. Acute pancreatitis. J Hosp Med. 2010 Apr;5(4):241-50. doi: 10.1002/jhm.574. PMID 20394032
- [Background] Raimondi S, Maisonneuve P, Lowenfels AB. Epidemiology of pancreatic cancer: an overview. Nat Rev Gastroenterol Hepatol. 2009 Dec;6(12):699-708. doi: 10.1038/nrgastro.2009.177. Epub 2009 Oct 6. PMID 19806144
- [Background] Satoh K, Shimosegawa T, Masamune A, Hirota M, Kikuta K, Kihara Y, Kuriyama S, Tsuji I, Satoh A, Hamada S; Research Committee of Intractable Diseases of the Pancreas. Nationwide epidemiological survey of acute pancreatitis in Japan. Pancreas. 2011 May;40(4):503-7. doi: 10.1097/MPA.0b013e318214812b. PMID 21499203
- [Background] Schreyer AG, Jung M, Riemann JF, Niessen C, Pregler B, Grenacher L, Hoffmeister A; German Society of Digestive and Metabolic Diseases (DGVS). S3 guideline for chronic pancreatitis - diagnosis, classification and therapy for the radiologist. Rofo. 2014 Nov;186(11):1002-8. doi: 10.1055/s-0034-1385005. Epub 2014 Aug 14. PMID 25122174
- [Background] Soliman AS, Zhang Q, Saleh T, Zarzour A, Selim M, Abdel-Fattah M, Abbruzzese JL. Pancreatic cancer mortality in Egypt: comparison to the United States pancreatic cancer mortality rates. Cancer Detect Prev. 2006;30(5):473-9. doi: 10.1016/j.cdp.2006.06.006. Epub 2006 Oct 25. PMID 17067749
- [Background] Stevens T, Lopez R, Adler DG, Al-Haddad MA, Conway J, Dewitt JM, Forsmark CE, Kahaleh M, Lee LS, Levy MJ, Mishra G, Piraka CR, Papachristou GI, Shah RJ, Topazian MD, Vargo JJ, Vela SA. Multicenter comparison of the interobserver agreement of standard EUS scoring and Rosemont classification scoring for diagnosis of chronic pancreatitis. Gastrointest Endosc. 2010 Mar;71(3):519-26. doi: 10.1016/j.gie.2009.10.043. PMID 20189510
- [Background] van Santvoort HC, Bakker OJ, Bollen TL, Besselink MG, Ahmed Ali U, Schrijver AM, Boermeester MA, van Goor H, Dejong CH, van Eijck CH, van Ramshorst B, Schaapherder AF, van der Harst E, Hofker S, Nieuwenhuijs VB, Brink MA, Kruyt PM, Manusama ER, van der Schelling GP, Karsten T, Hesselink EJ, van Laarhoven CJ, Rosman C, Bosscha K, de Wit RJ, Houdijk AP, Cuesta MA, Wahab PJ, Gooszen HG; Dutch Pancreatitis Study Group. A conservative and minimally invasive approach to necrotizing pancreatitis improves outcome. Gastroenterology. 2011 Oct;141(4):1254-63. doi: 10.1053/j.gastro.2011.06.073. Epub 2011 Jul 8. PMID 21741922
- [Background] Xiao AY, Tan ML, Wu LM, Asrani VM, Windsor JA, Yadav D, Petrov MS. Global incidence and mortality of pancreatic diseases: a systematic review, meta-analysis, and meta-regression of population-based cohort studies. Lancet Gastroenterol Hepatol. 2016 Sep;1(1):45-55. doi: 10.1016/S2468-1253(16)30004-8. Epub 2016 Jun 28. PMID 28404111
- [Background] Yadav D, Timmons L, Benson JT, Dierkhising RA, Chari ST. Incidence, prevalence, and survival of chronic pancreatitis: a population-based study. Am J Gastroenterol. 2011 Dec;106(12):2192-9. doi: 10.1038/ajg.2011.328. Epub 2011 Sep 27. PMID 21946280
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135